CLINICAL TRIAL: NCT07268976
Title: Effect of Jackfruit Consumption on Adipokine, Cerebral Response, Cognitive Performance and Anthropometric Parameters in Boxers
Brief Title: Jackfruit Effects on Adipokines and Cognition in Boxers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayburt University (Other)
Responsible Party: Principal Investigator, HATİCE BUDAK, Researcher / Principal Investigator/ Master's Student, Bayburt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BU-2025-01
Record Dates: First submitted 2025-08-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Exercise Physiology; Cognitive Function; Adipokine Response; Brain-Derived Neurotrophic Factor (BDNF); Irisin; Omentin-1
Keywords: Boxer; Athletes; Jackfruit; Irisin; Omentin-1; BDNF; Cognitive Performance; Anthropometric Measurements; Adipokines; Trail Making Test; Wisconsin Card Sorting Test (WCST); Body Composition

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to four parallel groups (J0, J100, J200, J300) receiving different doses of jackfruit oil extract (0, 100, 200, 300 mg/kg). Each group received the assigned intervention for 30 days, and outcomes including salivary irisin, omentin-1, BDNF levels, cognitive performance, and anthropometric measurements were assessed at baseline and at the end of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- J0 - Kontrol Grubu (No Intervention): Katılımcılar hiçbir jackfruit yağı ekstresi almadı. Sadece normal diyet ve antrenman programlarını sürdürdüler.
- J100 (Experimental): Katılımcılara 100 mg/kg jackfruit yağı ekstresi oral olarak 500 ml su içinde verildi. Müdahale 30 gün boyunca günlük olarak uygulandı.
  Interventions: Dietary Supplement: Jackfruit Supplement
- J200 (Experimental): Katılımcılara 200 mg/kg jackfruit yağı ekstresi oral olarak 500 ml su içinde verildi. Müdahale 30 gün boyunca günlük olarak uygulandı.
  Interventions: Dietary Supplement: Jackfruit Supplement
- J300 (Experimental): Katılımcılara 300 mg/kg jackfruit yağı ekstresi oral olarak 500 ml su içinde verildi. Müdahale 30 gün boyunca günlük olarak uygulandı.
  Interventions: Dietary Supplement: Jackfruit Supplement

INTERVENTIONS:
Dietary Supplement: Jackfruit Supplement — Participants in the experimental group will receive a daily dose of jackfruit supplement during the study period. The supplement is administered orally and standardized for bioactive components. Participants in the control group will not receive any jackfruit supplement.
  Arms: J100; J200; J300

SUMMARY:
This study investigates the effects of jackfruit oil extract on adipokine levels (Irisin, Omentin-1), brain-derived neurotrophic factor (BDNF), cognitive performance, and body measurements in healthy young boxers aged 18-25. Participants were randomly assigned to four groups receiving different doses of jackfruit oil extract (0, 100, 200, 300 mg/kg) or no supplement. Saliva samples, cognitive tests, and body measurements were collected at the start of the study and after 30 days to evaluate the outcomes.

DETAILED DESCRIPTION:
This interventional study evaluates the effects of different doses of jackfruit oil extract on healthy young boxers aged 18-25. Participants were randomly assigned to four groups and followed for 30 days.

Saliva samples were collected to measure irisin, omentin-1, and BDNF levels. Cognitive performance was assessed using the Wisconsin Card Sorting Test and the Trail Making Test. Anthropometric parameters including weight, BMI, waist, hip, chest, limb circumferences, and body composition were measured at baseline and on day 30.

Statistical analyses were performed using SPSS version 26. ANOVA, Duncan, and Pearson correlation tests were used to determine significant differences and relationships between variables.

This study is randomized and controlled. Participants receive either one of three doses of jackfruit oil extract or no supplement. The follow-up period is 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Male boxers aged 18-25 years
* Healthy individuals without any diagnosed chronic disease
* Participating in regular weekly boxing training
* Able to continue training throughout the study period
* Willing to voluntarily participate in the study
* Able to provide written and/or verbal informed consent

Exclusion Criteria:

* Presence of chronic diseases (e.g., diabetes, cardiovascular disorders)
* Any injury or musculoskeletal condition preventing continuation of training
* Known allergy or hypersensitivity to jackfruit or its components
* Use of medications or supplements that could interfere with study outcomes
* Individuals who refuse to provide informed consent

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Salivary Irisin Level | Day 0 and Day 30
  Irisin levels measured from saliva samples collected from participants using the ELISA method.
Salivary Omentin-1 Level | Day 0 and Day 30.
  Omentin-1 levels measured from saliva samples collected from participants using the ELISA method.
Salivary BDNF Level | Day 0 and Day 30.
  BDNF levels measured from saliva samples collected from participants using the ELISA method.

SECONDARY OUTCOMES:
Body Weight (kg) | Day 0 and Day 30
  Body weight measured using Tanita BC-418 bioimpedance device.
Height (cm) | Day 0 and Day 30
  Height measured using a standard stadiometer.
Body Mass Index (kg/m²) | Day 0 and Day 30
  BMI calculated using the formula weight (kg)/height (m²).
Waist Circumference (cm) | Day 0 and Day 30
  Waist circumference measured with a flexible tape measure.
Hip Circumference (cm) | Day 0 and Day 30
  Hip circumference measured with a flexible tape measure.
Chest Circumference (cm) | Day 0 and Day 30
  Chest circumference measured using a flexible tape measure.
Upper Arm Circumference (Right/Left, cm) | Day 0 and Day 30
  Right and left upper arm circumferences measured with a flexible tape measure.
Wrist Circumference (Right/Left, cm) | Day 0 and Day 30
  Right and left wrist circumferences measured with a flexible tape measure.
Thigh Circumference (Right/Left, cm) | Day 0 and Day 30
  Right and left thigh circumferences measured with a flexible tape measure.
Calf Circumference (Right/Left, cm) | Day 0 and Day 30
  Right and left calf circumferences measured with a flexible tape measure.
Total Body Fat Mass (kg) | Day 0 and Day 30
  Total body fat mass measured using Tanita BC-418.
Total Body Fat Percentage (%) | Day 0 and Day 30
  Total body fat percentage measured using Tanita BC-418.
Abdominal Fat Mass (kg) | Day 0 and Day 30
  Abdominal fat mass measured using Tanita BC-418.
Regional Fat Percentages (Right/Left Arm & Leg) | Day 0 and Day 30
  Regional fat percentages for arms and legs measured by Tanita BC-418.
Total Muscle Mass (kg) | Day 0 and Day 30
  Total muscle mass assessed using Tanita BC-418.
Regional Muscle Mass (Right/Left Arm & Leg, kg) | Day 0 and Day 30
  Regional muscle mass of arms and legs measured by Tanita BC-418.
Basal Metabolic Rate (BMR) | Day 0 and Day 30
  Basal metabolic rate calculated by Tanita BC-418.
Metabolic Age | Day 0 and Day 30
  Metabolic age estimated using Tanita BC-418 device.
Total Body Water (kg) | Day 0 and Day 30
  Total body water measured via bioimpedance analysis.
Total Body Water Percentage (%) | Day 0 and Day 30
  Total Body Water Percentage (%)
WCST Total Correct Responses | Day 0 and Day 30
  Total correct responses obtained from the Wisconsin Card Sorting Test.
WCST Total Incorrect Responses | Day 0 and Day 30
  Total incorrect responses measured using the Wisconsin Card Sorting Test.
WCST Perseverative Error Count | Day 0 and Day 30
  Perseverative errors recorded during the Wisconsin Card Sorting Test.
WCST Total Time (seconds) | Day 0 and Day 30
  Total time required to complete the Wisconsin Card Sorting Test.
Trail Making Test A Completion Time (seconds) | Day 0 and Day 30
  Completion time for Trail Making Test Part A.
Trail Making Test B Completion Time (seconds) | Day 0 and Day 30
  Completion time for Trail Making Test Part B.
Biomarker Correlations (Irisin-Omentin-BDNF vs. Dose/Day) | Based on Day 30 measurements
  Pearson correlation analysis examining relationships between biomarkers and intervention dose/day.
Safety Outcomes (Adverse Event Monitoring) | Continuous monitoring throughout 30 days
  Monitoring of potential adverse events related to 300 mg/kg JOE administration.

CONTACTS AND LOCATIONS:
Overall Officials: BÜLENT BAYRAKTAR, Principal Investigator — BAYBURT ÜNİVERSİTESİ
Locations (1):
- Bayburt Gençlik Merkezi Kapali Spor Salonu, Bayburt, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data including salivary irisin, omentin-1, BDNF levels, anthropometric measurements, and cognitive test results will be shared with other researchers upon reasonable request after publication of the main study results. Access will require approval from the institutional ethics committee and signing a data use agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified participant-level data and supporting documents will be available to other researchers starting after publication of the main study results and will remain accessible for 5 years following publication.
Access Criteria: "Access to de-identified participant-level data and supporting documents will be granted to qualified researchers for legitimate scientific purposes. Researchers must submit a request detailing their research objectives and methods, obtain approval from the institutional ethics committee, and sign a data use agreement. Approved researchers will receive access to the specified datasets and supporting materials electronically.
URL: https://www.bayburt.edu.tr/en/faculty-of-health-sciences/research

REFERENCES:
- See also: This study investigates the effects of jackfruit consumption on adipokine levels (irisin, omentin-1), brain-derived neurotrophic factor (BDNF), cognitive performance, and anthropometric parameters in young boxers aged 18-25. — https://www.bayburt.edu.tr/spor-bilimleri